CLINICAL TRIAL: NCT06823973
Title: Anthesis - A Transdiagnostic Approach to Sexual Distress: Testing a Pilot Online Intervention
Brief Title: Anthesis: A Transdiagnostic Cognitive-Behavioral Therapy (CBT)-Based Approach to Sexual Distress: Testing a Pilot Online Intervention
Acronym: Anthesis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo Lusófona (Other)
Responsible Party: Principal Investigator, Patrícia M. Pascoal, Professor, Grupo Lusófona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022.09087.PTDC; 2022.09087.PTDC (Other: Fundação para a Ciência e a Tecnologia)
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Sexual Distress; Sexual Dysfunctions
Keywords: Sexual distress related to sexual function; Sexual distress; Cognitive behavioural therapy; Transdiagnostic approach; Online intervention; Pilot study

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention condition (Experimental): Participants will access the treatment (Anthesis) by logging in to the platform. Each week, a new module is presented. During the week, participants can log onto the platform regularly to view each week's module, complete the homework presented at the end of each module, and proceed to the new module. Participants can contact the therapist through a written message during the intervention. All communication between the therapist and participants will occur exclusively through the platform.
  Interventions: Behavioral: CBT-based transdiagnostic approach to sexual distress
- Waiting list control condition (Other): The participants in the waiting list condition will not receive the intervention, while the participants in the experimental condition complete the protocol. However, participants in the waiting list condition have the option to contact the research team if their symptoms worsen or if they have any concerns related to the program. Once the participants in the experimental condition finish the intervention, the participants in the waiting list condition will then receive the intervention.
  Interventions: Behavioral: Waiting list condition

INTERVENTIONS:
Behavioral: CBT-based transdiagnostic approach to sexual distress — It is constituted by 8 modules:
  1. Psychoeducation about sexual function
  2. Difficulties in emotional regulation
  3. Non-judgmental emotional awareness
  4. Cognitive flexibility
  5. Worry and rumination
  6. Perfectionism
  7. Communication
  8. Summary
  Arms: Intervention condition
Behavioral: Waiting list condition — The participants in the waiting list condition will receive the intervention after the participants in the intervention condition.
  Arms: Waiting list control condition

SUMMARY:
This pilot study, named Anthesis, evaluates the preliminary efficacy of an online pilot study for sexual distress related to sexual function (SDRSF) in adults. Anthesis is theoretically anchored on a transdiagnostic CBT-based approach to SDRSF. The experience of sexual distress, especially sexual distress related to sexual function (SDRSF), is associated with poorer physical health, poorer mental health, and relational conflicts, which makes the development of theoretically and empirically sustained clinical interventions to eliminate or minimize it fundamental. In this project, the authors will attempt to answer the overall research question: "Does an online intervention aimed at transdiagnostic factors prove to have preliminary efficacy in reducing SDRSF?" Driven by both theory and empirical evidence on the comorbidity between emotional disorders and sexual dysfunctions, this project will focus on SDRSF (as a primary outcome variable). It will be considered a secondary outcome of sexual function and sexual pleasure.

Anthesis consists of eight modules (one module per week) delivered online. Participants will be divided into two conditions: an experimental condition that will start the intervention after the screening and a waiting list control condition (WLC) that will only begin its intervention after participants in the experimental condition have completed it.

DETAILED DESCRIPTION:
Background: According to DSM-5-TR and ICD-11, the experience of some level of sexual distress is an essential condition to establish a diagnosis of sexual dysfunction (SD). Recent research suggests high comorbidity between several clinical conditions and SD (e.g., between depression and decreased desire; between anxiety and orgasmic difficulties), as well as the presence of psychological processes (e.g., perfectionism, emotional dysregulation, worry) in the aetiology and maintenance of several SD. These processes are also common to other emotional disorders. This relation between vulnerability and maintenance factors of emotional disorders and SDs suggests that a transdiagnostic approach, which studies factors common to different emotional problems, will be adequate to intervene in SDRSF.

Research conducted worldwide indicates that most people facing distressing sexual problems do not actively seek or receive professional help. Many people feel ashamed to ask for health support for SDs and sexual problems. Additionally, various barriers-such as financial constraints, time limitations, long waiting lists, and a lack of specialists in sexual problems-hinder access to clinical support and negatively impact people's well-being and relationships. Therefore, the authors propose developing an online intervention that the literature indicates may increase accessibility to psychological interventions and help to overcome these barriers.

This project, focused on eliminating or reducing SDRSF, involves a pilot randomized controlled trial with participants divided into an intervention condition and a waiting list condition. Potential participants will be screened for eligibility using questionnaires to evaluate SDRSF, sexual function and general sexual distress on the intervention platform. After this, the eligibility criteria will be verified through screening during a clinical phone interview. Before starting the intervention, all participants will be informed about the study details on an informed consent form and will be given contact information from the research team for further clarification, if needed. The entire intervention will occur through a secure online platform. The Anthesis protocol aims to a) reduce sexual distress related to sexual function, b) improve sexual function, and c) increase sexual pleasure.

ELIGIBILITY:
The inclusion criteria are:

1. experiencing distress related to sexual function
2. understanding Portuguese
3. being over 18 years old
4. being in an exclusive (monogamic) romantic relationship for more than six months

Potential participants will be excluded if they are:

1. taking medication that interferes with the sexual response (e.g., antipsychotics, antidepressants, some types of hormone therapy or other)
2. having medical conditions that could impact the intervention outcomes (e.g., cancer, diabetes)
3. currently receiving psychological treatment, including psychological treatment for sexual dysfunctions or sexual problems
4. a transgender or intersex person
5. experiencing sexual pain

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Cisgender men Cisgender women
Enrollment: 30 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change from Sexual Function Evaluation Questionnaire | Baseline, post-intervention assessment (8 weeks after the baseline) and follow-up assessments at 3 months
  Sexual problems are assessed using the Sexual Function Evaluation Questionnaire (SFEQ), which includes 16 items divided into four factors: distress related to sexual function (factor 1), partner relationships (factor 2), overall sex life (factor 3), and sexual confidence (factor 4). Responses are based on individuals' experiences over the past month, with four different options available. Higher scores for Factors 1, 2, and 3, combined with lower scores for Factor 4, indicate poorer sexual function. In the overall evaluation, higher total scores also represent lower sexual function, with a minimum total score of 16 and a maximum total score of 64.

SECONDARY OUTCOMES:
Change from Sexual Distress Scale | Baseline, post-intervention assessment (8 weeks after the baseline) and follow-up assessments at 3 months
  Sexual distress is assessed using the Sexual Distress Scale (SDS), a unidimensional scale consisting of 12 items. Each item is evaluated on a Likert-type scale ranging from 0 to 4, with higher scores denoting increased sexual distress experienced over the past 30 days. The minimum score is 0, and the maximum total score is 48, with higher scores suggesting greater sexual distress.
Change from International Index of Erectile Function | Baseline, post-intervention assessment (8 weeks after the baseline) and follow-up assessments at 3 months
  Male sexual function is assessed using the International Index of Erectile Function (IIEF), which consists of 15 items distributed across five factors: erectile function (factor 1), orgasmic function (factor 2), sexual desire (factor 3), intercourse satisfaction (factor 4), and overall satisfaction (factor 5). Each item is rated on a Likert-type scale from 0 to 5-where lower scores indicate greater male sexual dysfunction experienced over the last four weeks. In instances where no sexual activity occurred, a score of 0 is given. The maximum total score is 75, with lower overall scores suggesting an increased risk of sexual dysfunction.
Change from Female Sexual Function Index | Baseline, post-intervention assessment (8 weeks after the baseline) and follow-up assessments at 3 months
  Female sexual function is measured using the Female Sexual Function Index (FSFI), which comprises 19 items distributed across six factors: desire (factor 1), arousal (factor 2), lubrication (factor 3), orgasm (factor 4), satisfaction (factor 5), and pain (factor 6). Each item is rated on a Likert-type scale ranging from 1 to 5-with lower scores indicating greater dysfunction over the past 4 weeks-and in cases where no sexual activity occurred, a score of 0 is assigned. The maximum total score is 36, with lower values suggesting a risk of sexual dysfunction.
Change from Sexual Pleasure Scale | Baseline, post-intervention assessment (8 weeks after the baseline) and follow-up assessments at 3 months
  Sexual pleasure derived from sexual relationships, activities, and intimacy is assessed using the Sexual Pleasure Scale (SPS), a unidimensional scale that comprises 13 items. Each item on the scale is rated using a Likert-type scale ranging from 0 to 4, with higher scores indicating greater sexual pleasure. The minimum total score is 0, which represents no sexual pleasure, while the maximum score is 52, indicating the highest level of sexual pleasure experienced.

CONTACTS AND LOCATIONS:
Locations (2):
- Portugal (2):
  - Lusófona University, Lisbon
  - Universidade Lusófona- Centro Universitário de Lisboa, Lisbon

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.

REFERENCES:
- [Background] Guerreiro, P. P., Raposo, C. F., Salvador, Á., Manão, A. A., & Pascoal, P. M. (2024). A transdiagnostic approach to sexual distress and pleasure: The role of worry, rumination, and emotional regulation. Current Psychology, 43(17), 15385-15396.
- [Background] American Psychiatric Association. (2022). Diagnostic and statistical manual of mental disorders (5th ed., text rev.). American Psychiatric Association. https://doi.org/10.1176/appi.books.9780890425787
- [Background] Tavares IM, Moura CV, Nobre PJ. The Role of Cognitive Processing Factors in Sexual Function and Dysfunction in Women and Men: A Systematic Review. Sex Med Rev. 2020 Jul;8(3):403-430. doi: 10.1016/j.sxmr.2020.03.002. Epub 2020 May 10. PMID 32402763
- [Background] Raposo CF, Nobre PJ, Manao AA, Pascoal PM. Understanding sexual distress related to sexual function (SDRSF): A preliminary framework based on a qualitative study with clinical sexologists. Int J Clin Health Psychol. 2024 Jul-Sep;24(3):100473. doi: 10.1016/j.ijchp.2024.100473. Epub 2024 Jun 24. PMID 39021678
- [Background] Quinta Gomes AL, Nobre P. Personality traits and psychopathology on male sexual dysfunction: an empirical study. J Sex Med. 2011 Feb;8(2):461-9. doi: 10.1111/j.1743-6109.2010.02092.x. Epub 2010 Nov 3. PMID 21054796
- [Background] Peixoto MM, Ribeiro V. Repetitive Negative Thinking and Sexual Functioning in Portuguese Men and Women: A Cross-Sectional Study. Int J Sex Health. 2022 Jun 7;34(4):567-576. doi: 10.1080/19317611.2022.2084201. eCollection 2022. PMID 38596387
- [Background] Pascoal PM, Raposo CF, Roberto MS. A Transdiagnostic Approach to Sexual Distress and Sexual Pleasure: A Preliminary Mediation Study with Repetitive Negative Thinking. Int J Environ Res Public Health. 2020 Oct 27;17(21):7864. doi: 10.3390/ijerph17217864. PMID 33121015
- [Background] Martins EM, Pascoal PM, Manao AA, Rosa PJ. The Interplay of Worry and Relationship Satisfaction to Understand Sexual Distress: An APIM Study with Heterosexual Couples Using Cross-Sectional Data. J Sex Marital Ther. 2024;50(7):878-893. doi: 10.1080/0092623X.2024.2391390. Epub 2024 Aug 26. PMID 39183638
- [Background] Manao AA, Martins E, Pascoal PM. What Sexual Problems Does a Sample of LGB+ People Report Having, and How Do They Define Sexual Pleasure: A Qualitative Study to Inform Clinical Practice. Healthcare (Basel). 2023 Oct 30;11(21):2856. doi: 10.3390/healthcare11212856. PMID 37958001
- [Background] Manao AA, Pascoal PM. Body Dissatisfaction, Cognitive Distraction, and Sexual Satisfaction in a Sample of LGB+ People: A Mediation Study Framed by Cognitive Psychology Models of Sexual Response. Healthcare (Basel). 2023 Nov 9;11(22):2930. doi: 10.3390/healthcare11222930. PMID 37998422
- [Background] Hendrickx L, Gijs L, Enzlin P. Distress, sexual dysfunctions, and DSM: dialogue at cross purposes? J Sex Med. 2013 Mar;10(3):630-41. doi: 10.1111/j.1743-6109.2012.02971.x. Epub 2012 Oct 22. PMID 23088564
- [Background] Hayes RD, Dennerstein L, Bennett CM, Sidat M, Gurrin LC, Fairley CK. Risk factors for female sexual dysfunction in the general population: exploring factors associated with low sexual function and sexual distress. J Sex Med. 2008 Jul;5(7):1681-93. doi: 10.1111/j.1743-6109.2008.00838.x. PMID 18410300
- [Background] Costa IB, Manao AA, Pascoal PM. Clinical Sexologists' Perceptions of the Potentials, Downfalls, and Best Practices for Digitally Delivered Therapy: A Lesson from Lockdown Due to COVID-19 in Portugal. Behav Sci (Basel). 2023 May 4;13(5):376. doi: 10.3390/bs13050376. PMID 37232613
- [Background] Carvalho J, Nobre P. Predictors of women's sexual desire: the role of psychopathology, cognitive-emotional determinants, relationship dimensions, and medical factors. J Sex Med. 2010 Feb;7(2 Pt 2):928-37. doi: 10.1111/j.1743-6109.2009.01568.x. Epub 2009 Nov 13. PMID 19912503
- [Background] Brotto LA, Atallah S, Carvalho J, Gordon E, Pascoal PM, Reda M, Stephenson KR, Tavares IM. Psychological and interpersonal dimensions of sexual function and dysfunction: recommendations from the fifth international consultation on sexual medicine (ICSM 2024). Sex Med Rev. 2025 Apr 14;13(2):118-143. doi: 10.1093/sxmrev/qeae073. PMID 39786497
- [Background] Beato AF, Pascoal PM, Rodrigues J. The impact of digital media on sexuality: a descriptive and qualitative study. Int J Impot Res. 2024 Nov;36(7):770-780. doi: 10.1038/s41443-024-00865-y. Epub 2024 Mar 14. PMID 38486121